CLINICAL TRIAL: NCT02102334
Title: Validity, Reliability and Reproducibility of Plain Radiographic Measurements After Total Hip Arthroplasty
Status: Completed | Type: Observational
Sponsor: Sundsvall Hospital (Other)
Responsible Party: Principal Investigator, Lennart Bråbäck, MD, PhD, Sundsvall Hospital
Other Study IDs: RMVL
Record Dates: First submitted 2014-03-29; First posted 2014-04-02 (Estimated); Last update posted 2014-04-02 (Estimated); Status verified 2014-03

CONDITIONS: Osteoarthritis of the Hip
Keywords: Osteoarthritis, hip,; radiograpghic measurements; femoral offset; leg length discrepancy; cup anteversion; cup inclination
MeSH Terms: conditions — Osteoarthritis, Hip; Leg Length Inequality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Unilateral osteoarthritis: Patients operated with a total hip replacement due to unilateral osteoarthritis of the hip. Radiographic measurements of the postoperative radiographs.

SUMMARY:
In total hip arthroplasty (THA), radiographic preoperative planning and postoperative evaluation of acetabular component, femoral offset (FO) and leg length discrepancy (LLD) require good validity, interobserver reliability and intraobserver reproducibility.

Questions/purposes: (1) Evaluate the validity of the Sundsvall method of FO measurement by comparing it to a standard FO measurement method. (2) Evaluate the interobserver reliability and intraobserver reproducibility of measurement of FO, LLD, acetabular cup inclination and anteversion.

90 patients with primary unilateral osteoarthritis (OA) were included in this prospective study. On postoperative radiographs FO by the Sundsvall method, FO by a standard method, LLD, acetabular cup inclination and anteversion were measured. The interobserver reliability and intraobserver reproducibility were made by three independent observers. The validity and degree of prediction of Sundsvall method are measured by comparing its results with the standard method.

ELIGIBILITY:
Inclusion Criteria:

* unilateral total hip replacement with either a cemented Lubinus SP II system (Link, Germany) or an uncemented CLS stem and Triology cup (Zimmer, U.S.A).

Exclusion Criteria:

* Patient with secondary (OA), previous spinal, pelvic, or lower limb injuries or fractures were excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 90 consecutive patients with primary unilateral osteoarthritis (OA) who underwent THA between September 2010 and June 2012 were recruited into the study.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2010-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Leg Length Discrepancy | 1 week
  LLD on radiographs was defined as the difference in perpendicular distance in millimetres between a line passing through the lower edge of the teardrop points to the corresponding tip of the lesser trochanter. The interobserver reliability was assessed from the measurements made by three independent observers.
Femoral offset (Sundsvall method) | 1 week
  Measurement of FO using the Sundsvall method was carried out on the AP view of the pelvis as the horizontal distance (parallel to Hilgenreiners line) between the femoral axis (a line drawn through the center of the femoral shaft) and the mid line of the pelvis, at the height of the lateral tip of the greater trochanter. The measurement was performed bilaterally to compare the femoral offset on the operated side to the non-operated hip. The interobserver reliability was assessed from the measurements made by three independent observers.
Femoral offset (standard method) | 1 week
  Measurement of FO with the standard method was carried out on AP view as the addition of the distance between the longitudinal axis of the femur to center of femoral head and the distance from the center of the femoral head to a perpendicular line passing through the medial edge of the ipsilateral teardrop point of the pelvis. The measurement was repeated bilaterally to compare the FO of the operated side to non-operated hip. The interobserver reliability was assessed from the measurements made by three independent observers.
Cup inclination | 1 week
  Cup inclination was measured on AP view as angle in degrees, between a line drawn along the angle of rim of the cup and trans-ischial line (a line drawn between the most inferior point of the ischial tuberosities). The interobserver reliability was assessed from the measurements made by three independent observers.
Acetabular cup anteversion | 1 week
  Acetabular cup anteversion was measured on lateral radiograph as the angle formed by the intersection of a line drawn across the face of acetabulum and a line perpendicular to the horizontal plane, according to the Woo and Morry method. The interobserver reliability was assessed from the measurements made by three independent observers.

CONTACTS AND LOCATIONS:
Overall Officials: Arkan S Sayed-Noor, MD,PhD,FRCS, Principal Investigator — Umeå University
Locations (1):
- Sundsvall hostpital, Sundsvall, Västernorrland County, Sweden

REFERENCES:
- [Background] Kjellberg M, Englund E, Sayed-Noor AS. A new radiographic method of measuring femoral offset. The Sundsvall method. Hip Int. 2009 Oct-Dec;19(4):377-81. doi: 10.1177/112070000901900413. PMID 20041386
- [Background] Lecerf G, Fessy MH, Philippot R, Massin P, Giraud F, Flecher X, Girard J, Mertl P, Marchetti E, Stindel E. Femoral offset: anatomical concept, definition, assessment, implications for preoperative templating and hip arthroplasty. Orthop Traumatol Surg Res. 2009 May;95(3):210-9. doi: 10.1016/j.otsr.2009.03.010. Epub 2009 May 6. PMID 19423418
- [Background] Gililland JM, Anderson LA, Boffeli SL, Pelt CE, Peters CL, Kubiak EN. A fluoroscopic grid in supine total hip arthroplasty: improving cup position, limb length, and hip offset. J Arthroplasty. 2012 Sep;27(8 Suppl):111-6. doi: 10.1016/j.arth.2012.03.027. Epub 2012 May 3. PMID 22560563
- [Background] Konyves A, Bannister GC. The importance of leg length discrepancy after total hip arthroplasty. J Bone Joint Surg Br. 2005 Feb;87(2):155-7. doi: 10.1302/0301-620x.87b2.14878. PMID 15736733
- [Background] Bonett DG. Sample size requirements for estimating intraclass correlations with desired precision. Stat Med. 2002 May 15;21(9):1331-5. doi: 10.1002/sim.1108. PMID 12111881
- [Background] Woolson ST, Hartford JM, Sawyer A. Results of a method of leg-length equalization for patients undergoing primary total hip replacement. J Arthroplasty. 1999 Feb;14(2):159-64. doi: 10.1016/s0883-5403(99)90119-5. PMID 10065720
- [Background] Wylde V, Maclean A, Blom AW. Post-operative radiographic factors and patient-reported outcome after total hip replacement. Hip Int. 2012 Mar-Apr;22(2):153-9. doi: 10.5301/HIP.2012.9225. PMID 22547373
- [Background] Wylde V, Whitehouse SL, Taylor AH, Pattison GT, Bannister GC, Blom AW. Prevalence and functional impact of patient-perceived leg length discrepancy after hip replacement. Int Orthop. 2009 Aug;33(4):905-9. doi: 10.1007/s00264-008-0563-6. Epub 2008 Apr 25. PMID 18437379
- [Background] Little NJ, Busch CA, Gallagher JA, Rorabeck CH, Bourne RB. Acetabular polyethylene wear and acetabular inclination and femoral offset. Clin Orthop Relat Res. 2009 Nov;467(11):2895-900. doi: 10.1007/s11999-009-0845-3. Epub 2009 May 2. PMID 19412648
- [Background] Patel SR, Toms AP, Rehman JM, Wimhurst J. A reliability study of measurement tools available on standard picture archiving and communication system workstations for the evaluation of hip radiographs following arthroplasty. J Bone Joint Surg Am. 2011 Sep 21;93(18):1712-9. doi: 10.2106/JBJS.J.00709. PMID 21938375
- [Background] Kjellberg M, Al-Amiry B, Englund E, Sjoden GO, Sayed-Noor AS. Measurement of leg length discrepancy after total hip arthroplasty. The reliability of a plain radiographic method compared to CT-scanogram. Skeletal Radiol. 2012 Feb;41(2):187-91. doi: 10.1007/s00256-011-1166-7. Epub 2011 Apr 14. PMID 21491155
- [Background] Moskal JT, Capps SG. Acetabular component positioning in total hip arthroplasty: an evidence-based analysis. J Arthroplasty. 2011 Dec;26(8):1432-7. doi: 10.1016/j.arth.2010.11.011. Epub 2011 Feb 5. PMID 21296551